CLINICAL TRIAL: NCT05976126
Title: Characterization of a Population Living in Highly Contaminated Settlement in Campania Region
Acronym: SPES
Status: Completed | Type: Observational
Sponsor: Francesca De Filippis (Other)
Responsible Party: Sponsor-Investigator, Francesca De Filippis, Professor, Federico II University
Organization: Federico II University (Other)
Other Study IDs: 59
Record Dates: First submitted 2023-07-20; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Environmental-Pollution-Related Condition
Keywords: dioxins; persistent organic pollutants; heavy metals; gut microbiome
MeSH Terms: interventions — Polychlorinated Biphenyls; Trace Elements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fecal samples were self-collected and frozen at -80°C for microbial DNA extraction; peripheral blood (about 100 mL in several aliquots) was collected from the volunteers, in the early morning, in blood collection tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High environmental pollution group (HIGH): subjects living in area characterized by high environmental pollution, as defined by Pizzolante et al. [Development of a municipality index of environmental pressure in Campania, Italy. Future Sci. OA 7(7), FSO720 (2021).]
  Interventions: Other: Determination of dioxins (PCDD/Fs), polychlorinated biphenyls (PCBs) and trace elements
- Medium environmental pollution group (MEDIUM): subjects living in area characterized by medium environmental pollution, as defined by Pizzolante et al. [Development of a municipality index of environmental pressure in Campania, Italy. Future Sci. OA 7(7), FSO720 (2021).]
  Interventions: Other: Determination of dioxins (PCDD/Fs), polychlorinated biphenyls (PCBs) and trace elements
- Low environmental pollution group (LOW): subjects living in area characterized by low environmental pollution, as defined by Pizzolante et al. [Development of a municipality index of environmental pressure in Campania, Italy. Future Sci. OA 7(7), FSO720 (2021).]
  Interventions: Other: Determination of dioxins (PCDD/Fs), polychlorinated biphenyls (PCBs) and trace elements

INTERVENTIONS:
Other: Determination of dioxins (PCDD/Fs), polychlorinated biphenyls (PCBs) and trace elements — Peripheral blood (about 100 mL in several aliquots) was collected from the volunteers, in the early morning, in blood collection tubes (SST II Advance Tubes, BD Vacutainer). The samples were left for approximately 50 min, then the serum was separated from whole blood by centrifugation at 2,000 rcf for 10 min at 4 °C and then aliquots were stored at -80°C until analysis.

SUMMARY:
some areas in the Campania region (southern Italy) have attracted media coverage in the past 15 years, and are considered a dramatic example of an extremely polluted area. The environmental pollution issue has become a significant concern in the Campania Region as a result of the "waste management crisis" that mainly affects the northern part of the region, encompassing 91 municipalities. As a consequence, in the last few decades, a large rural area between the provinces of Naples and Caserta, primarily used for agriculture and livestock breeding, was considered to be at high risk of contamination due to the illegal disposal of urban and industrial waste. In these landfills, a broad range of hazardous wastes from different parts of Italy has been found. In addition, the wastes have often been open-air burned, leading to this area being named the "Land of Fires". Senior and Mazza first highlighted the high incidence of cancer deaths in a specific area of the Campania region (compared to regional and national rates), which was identified by the authors as the "triangle of death". Afterwards, several studies reported a link between illegal waste disposal and an increased risk of cancer for the population, potentially associated with human exposure to carcinogenic substances such as dioxins, dioxin-like compounds, or polycyclic aromatic hydrocarbons, which can be released into air, soil, and water bodies through the illegal dumping and burning of waste. Within this study, 4,227 subjects were enrolled in the SPES trial, considering healthy subjects living in several regional areas with different environmental pressures. Blood dioxins and heavy metals were analyzed. Gut microbiome was analyzed on a subset of 359 subjects from the three different exposure area.

DETAILED DESCRIPTION:
This study involved a screening of healthy adults from Campania region recruited in the human biomonitoring study SPES (http://spes.campaniatrasparente.it), promoted by the Istituto Zooprofilattico Sperimentale del Mezzogiorno (IZSM) of Portici (Italy) in collaboration with the National Tumor Institute IRCCS (Istituto di Ricovero e Cura a Carattere Scientifico) "G. Pascale" in Naples. Considering different source of environmental pressure (e.g., land use and population density, presence of contaminated sites, quality of air, soil and water bodies, closeness to waste management plants and illegal waste spills and fires), Pizzolante and colleagues developed an integrated model to compute the Municipality Index of Environmental Pressure (MIEP). The MIEP takes into account all factors involved in the pollution processes, including the sources of contaminants and their migration pathways. The MIEP enables the identification of 21 homogeneous sub-clusters, which include several municipalities based on their environmental pressure scores. This categorization has resulted in three macro-areas with increasing levels of impact pressure: LOW, MEDIUM and HIGH, as described by Pierri and colleagues. In 2016, a total of 4,227 subjects were enrolled in the SPES trial, considering healthy subjects living in several regional areas with different environmental pressures. A subgroup of 359 subjects residing in the three impact areas was randomly selected from the entire SPES cohort for gut microbiome analysis, in order to define the impact of environmental pollution on gut microbial communities.

ELIGIBILITY:
Inclusion criteria:

* healthy subjects (no severe, chronic or neoplastic conditions)
* 20-50 years old
* both sexes
* no important viral infection (HIV, HCV, HBV)
* no use of drugs
* no alcohol abuse
* no obesity of II, III and IV classes.
* resident in one of the municipalities under study for at least 5 years (Campania Region, Italy)

Exclusion criteria:

* age < 20 and > 50 years at enrollment
* severe, chronic or neoplastic conditions
* viral infections (HIV, HCV, HBV)
* use of drugs or alcohol
* obesity

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults (20-50 years/old) resident in one of the municipalities under study for at least 5 years (Campania Region, Italy) grouped according to the environmental impact (high, medium and low) (as reported in http://www.campaniatrasparente.it)
Sampling Method: Non-Probability Sample
Enrollment: 4227 (Actual)
Dates: Start 2016-09-10 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Comparison of plasmatic concentration of dioxins (PCDD/Fs) and polychlorinated biphenyls (PCBs) in subjects from high, medium and low pollution area as assessed by HRGC-HRMS | at enrollement
  measure of PCDD/Fs and PCBs in human blood serum using High-Resolution Gas Chromathography coupled to High-Resolution Mass Spectrometry (HRGC-HRMS) analysis
Comparison of plasmatic concentration of trace elements in subjects from high, medium and low pollution area as assessed by ICP-MS | at enrollement
  trace elements (arsenic, beryllium, cadmium, cobalt, chromium, copper, iron, mercury, lithium, manganese, molybdenum, nickel, lead, antimony, selenium, strontium, thallium, vanadium, and zinc) were determined in human plasma using an inductively coupled plasma mass spectrometer (ICP-MS)
Comparison of gut microbiome composition and functions in subjects from high, medium and low pollution area as assessed by metagenomics | at enrollement
  Microbiome composition and potential functions was determined by shotgun metagenomics (Illumina paired-end sequencing, 2x150bp). The massive amount of sequences obtained was analyzed by using state of the art bioinformatics tools and the presence and relative abundance of the microbial species and genes occurring in each sample was determined.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Filippis F, Valentino V, Sequino G, Borriello G, Riccardi MG, Pierri B, Cerino P, Pizzolante A, Pasolli E, Esposito M, Limone A, Ercolini D. Exposure to environmental pollutants selects for xenobiotic-degrading functions in the human gut microbiome. Nat Commun. 2024 May 27;15(1):4482. doi: 10.1038/s41467-024-48739-7. PMID 38802370